CLINICAL TRIAL: NCT04242784
Title: IMPlementation of Best PRactices fOr Acute Stroke Care - Developing and Optimizing Regional Systems of Stroke Care
Brief Title: IMPROVE Stroke Care- Developing and Optimizing Regional Systems of Stroke Care
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry); Daiichi Sankyo (Industry); Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00076593
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Acute Stroke; Intracranial Hemorrhages; Subarachnoid Hemorrhage
MeSH Terms: conditions — Stroke; Intracranial Hemorrhages; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Spoke Hospital: Patients that undergo the Code Stroke process at Spoke Hospitals
- Hub Hospital: Patients that undergo the Code Stroke process at Hub Hospitals
- Transfer: Patients that undergo the Code Stroke process at a Spoke Hospital and transfer to the Hub Hospital

SUMMARY:
The purpose of this program is to develop a regional integrated stroke system that identifies, classifies, and treats patients with acute ischemic stroke more rapidly and effectively with reperfusion therapy.

DETAILED DESCRIPTION:
The design is based upon the implementation of best practice, that is, based on a comprehensive review of AHA guidelines regarding treatment of acute stroke, ICH (intracranial hemorrhage) and SAH(sub arachnoid hemorrhage). In the second phase, the project will be doing national and international surveys of best practices among comprehensive stroke centers and then combine evidence based guidelines and recommendation as well as expert consensus and guidelines when high level evidence is not available from the published literature. The aim to improve public stroke awareness, stroke symptom recognition within the time benefit window for treatment and calling 9-1-1, EMS transportation, and the proportion and speed of reperfusion therapy (fibrinolytic and in appropriate patients- endovascular treatment) in eligible patients. These improvements in acute stroke care delivery are expected to result in lower mortality, fewer recurrent strokes, and improved long term functional outcomes that we will measure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age who undergo the local acute code stroke process

Exclusion Criteria:

* In house patients with stroke are not included in this data set.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo the Acute Code Stroke Process, who demonstrate symptoms of a possible acute stroke, and are presenting to a Spoke or Hub within the Southeastern US at the 9 Hub Hospitals and Spokes associated with those Hubs participating in the project.
Sampling Method: Non-Probability Sample
Enrollment: 21646 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Time from door to drug as measured by medical record | From baseline (Q1, 2017), to Quarter 4 (2020)
  The time frame starting from the earliest time that the patient is documented as arriving to the hospital to the beginning time of the administration of the drug (TPA)
Change in Time from Door to Tici 2c/3 flow measured by medical record | From baseline (Q1, 2017), to Quarter 4 (2020)
  The time frame starting from the earliest time that the patient is documented as arriving to the hospital to the beginning time of Tici 2c/c flow noted in the vessel
Change in Time from Door to Administration of Reversal Agent as measured by medical record | From baseline (Q1, 2017), to Quarter 4 (2020)
  The time frame starting from the earliest time that the patient is documented as arriving to the hospital to the beginning time of the administration of the drug (reversal agent)

SECONDARY OUTCOMES:
Change in Number of Deaths from Stroke as measure by medical record | From baseline (Q1, 2017) to Quarter 4 (2020)
  Count of number of deaths from stroke
Change in Functional Long Term Outcomes as measured by Modified Rankin Scale | From baseline , 3 months
  Modified Ranking Scale ranges from 0-6,
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Graffagnino, MD, Principal Investigator — Duke University; Bradley Kolls, MD, Principal Investigator — Duke University
Locations (9):
- United States (9):
  - Mission Health, Asheville, North Carolina
  - Atrium Health's Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Prisma Health, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fonarow GC, Smith EE, Saver JL, Reeves MJ, Hernandez AF, Peterson ED, Sacco RL, Schwamm LH. Improving door-to-needle times in acute ischemic stroke: the design and rationale for the American Heart Association/American Stroke Association's Target: Stroke initiative. Stroke. 2011 Oct;42(10):2983-9. doi: 10.1161/STROKEAHA.111.621342. Epub 2011 Sep 1. PMID 21885841
- [Result] Fonarow GC, Zhao X, Smith EE, Saver JL, Reeves MJ, Bhatt DL, Xian Y, Hernandez AF, Peterson ED, Schwamm LH. Door-to-needle times for tissue plasminogen activator administration and clinical outcomes in acute ischemic stroke before and after a quality improvement initiative. JAMA. 2014 Apr 23-30;311(16):1632-40. doi: 10.1001/jama.2014.3203. PMID 24756513
- [Result] Xian Y, Xu H, Lytle B, Blevins J, Peterson ED, Hernandez AF, Smith EE, Saver JL, Messe SR, Paulsen M, Suter RE, Reeves MJ, Jauch EC, Schwamm LH, Fonarow GC. Use of Strategies to Improve Door-to-Needle Times With Tissue-Type Plasminogen Activator in Acute Ischemic Stroke in Clinical Practice: Findings from Target: Stroke. Circ Cardiovasc Qual Outcomes. 2017 Jan;10(1):e003227. doi: 10.1161/CIRCOUTCOMES.116.003227. PMID 28096207
- [Result] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Result] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Result] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Result] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Result] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Result] Powers WJ, Derdeyn CP, Biller J, Coffey CS, Hoh BL, Jauch EC, Johnston KC, Johnston SC, Khalessi AA, Kidwell CS, Meschia JF, Ovbiagele B, Yavagal DR; American Heart Association Stroke Council. 2015 American Heart Association/American Stroke Association Focused Update of the 2013 Guidelines for the Early Management of Patients With Acute Ischemic Stroke Regarding Endovascular Treatment: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Oct;46(10):3020-35. doi: 10.1161/STR.0000000000000074. Epub 2015 Jun 29. PMID 26123479
- [Result] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Result] Mellor RM, Bailey S, Sheppard J, Carr P, Quinn T, Boyal A, Sandler D, Sims DG, Mant J, Greenfield S, McManus RJ. Decisions and delays within stroke patients' route to the hospital: a qualitative study. Ann Emerg Med. 2015 Mar;65(3):279-287.e3. doi: 10.1016/j.annemergmed.2014.10.018. Epub 2014 Nov 15. PMID 25455907
- [Result] Shin CN, An K, Sim J. Facilitators of and barriers to emergency medical service use by acute ischemic stroke patients: A retrospective survey. Int J Nurs Sci. 2016 Dec 26;4(1):52-57. doi: 10.1016/j.ijnss.2016.12.008. eCollection 2017 Jan 10. PMID 31406718
- [Result] Ekundayo OJ, Saver JL, Fonarow GC, Schwamm LH, Xian Y, Zhao X, Hernandez AF, Peterson ED, Cheng EM. Patterns of emergency medical services use and its association with timely stroke treatment: findings from Get With the Guidelines-Stroke. Circ Cardiovasc Qual Outcomes. 2013 May 1;6(3):262-9. doi: 10.1161/CIRCOUTCOMES.113.000089. Epub 2013 Apr 29. PMID 23633218
- [Result] Schwamm LH, Audebert HJ, Amarenco P, Chumbler NR, Frankel MR, George MG, Gorelick PB, Horton KB, Kaste M, Lackland DT, Levine SR, Meyer BC, Meyers PM, Patterson V, Stranne SK, White CJ; American Heart Association Stroke Council; Council on Epidemiology and Prevention; Interdisciplinary Council on Peripheral Vascular Disease; Council on Cardiovascular Radiology and Intervention. Recommendations for the implementation of telemedicine within stroke systems of care: a policy statement from the American Heart Association. Stroke. 2009 Jul;40(7):2635-60. doi: 10.1161/STROKEAHA.109.192361. Epub 2009 May 7. No abstract available. PMID 19423851
- [Result] Wechsler LR, Demaerschalk BM, Schwamm LH, Adeoye OM, Audebert HJ, Fanale CV, Hess DC, Majersik JJ, Nystrom KV, Reeves MJ, Rosamond WD, Switzer JA; American Heart Association Stroke Council; Council on Epidemiology and Prevention; Council on Quality of Care and Outcomes Research. Telemedicine Quality and Outcomes in Stroke: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Jan;48(1):e3-e25. doi: 10.1161/STR.0000000000000114. Epub 2016 Nov 3. PMID 27811332
- [Result] Schulman S. Clinical practice. Care of patients receiving long-term anticoagulant therapy. N Engl J Med. 2003 Aug 14;349(7):675-83. doi: 10.1056/NEJMcp025373. No abstract available. PMID 12917305
- [Result] Aycock RD, Westafer LM, Boxen JL, Majlesi N, Schoenfeld EM, Bannuru RR. Acute Kidney Injury After Computed Tomography: A Meta-analysis. Ann Emerg Med. 2018 Jan;71(1):44-53.e4. doi: 10.1016/j.annemergmed.2017.06.041. Epub 2017 Aug 12. PMID 28811122